CLINICAL TRIAL: NCT03189914
Title: A Phase 1/2 Open-Label, Safety, Pharmacokinetic, Pharmacodynamic and Efficacy Study of RX-3117 in Combination With Abraxane® in Subjects With Metastatic Pancreatic Cancer
Brief Title: RX-3117 in Combination With Abraxane® in Subjects With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX3117-003
Record Dates: First submitted 2017-06-07; First posted 2017-06-16 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; Abraxane; first line
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — fluorocyclopentenylcytosine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RX-3117 + Abraxane (Experimental): RX-3117: oral, 500 - 700 mg/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 75 - 125 mg/m^2, infused once per week for 3 weeks. 1 washout week/ cycle.
  Interventions: Drug: RX-3117

INTERVENTIONS:
Drug: RX-3117 — RX-3117 will be administered orally in combination with Abraxane.
  Other Names: Abraxane

SUMMARY:
This will be a Phase 1b/2a multicenter 2-stage study. Phase 1 will be conducted as a dose-finding, open-label study of oral RX-3117 administered in combination with Abraxane® to subjects with metastatic pancreatic cancer. After completion of the Phase 1 portion, a Phase 2a study will be conducted using a 2 stage, open-label design, of RX 3117 and Abraxane® in combination to treat subjects with metastatic pancreatic cancer as first line therapy.

DETAILED DESCRIPTION:
This will be a Phase 1b/2a multicenter 2-stage study. Phase 1 will be conducted as a dose-finding, open-label study of oral RX-3117 administered in combination with Abraxane® to subjects with metastatic pancreatic cancer. The recommended phase 2 dose (RP2D) and schedule of RX-3117, in combination with Abraxane®, will be determined based on the safety profile, dose modification, and pharmacokinetics (PK). Phase 1 will be conducted using a combination of the single agent maximum tolerated dose (MTD) for RX-3117 and the Abraxane dose as per the package insert for patients with pancreatic cancer in combination with gemcitabine.

After completion of the Phase 1 portion, a Phase 2a study will be conducted using a 2 stage, open-label design, of RX 3117 and Abraxane® in combination to treat subjects with metastatic pancreatic cancer as first line therapy. Approximately 10 subjects will participate in the Stage 1 at the dose identified in Phase 1 (RP2D). Subjects will be treated for up to 8 cycles of combined therapy. An interim analysis will be conducted after 10 evaluable subjects have been treated at the RP2D, have completed a minimum of 4 cycles of therapy, or have discontinued therapy due to progressive disease before completing 4 cycles. If an adequate number of Responders are observed out of the initial 10 evaluable subjects, then 40 additional subjects will be enrolled to participate in Stage 2. Subjects will be treated for up to 8 cycles of combined therapy.

ELIGIBILITY:
Inclusion Criteria:

Disease Related

1. Subject has confirmed histologic or cytologic evidence of metastatic pancreatic cancer and has no prior treatment for metastatic pancreatic cancer.
2. Subject has measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
3. Subject has a life expectancy of at least 3 months.
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

   Demographic
5. Males or females ≥ 18 years of age
6. Subject must be able to swallow capsules
7. Subject must have adequate venous access for intravenous (IV) infusion

   Laboratory
8. Subject has hemoglobin ≥ 9.0 g/dL at Screening
9. Subject has absolute neutrophil count (ANC) ≥ 1.5 x 109/L at Screening
10. Subject has platelet count ≥ 100 x 109/L at Screening
11. Subject has serum creatinine ≤ 1.5 times the upper limit of normal (ULN) at Screening. Subjects with serum creatinine levels > 1.5 times the ULN must have a 24-hour urine creatinine clearance ≥ 60 mL/min
12. Subject has serum bilirubin ≤ 1.5 times the ULN (except in subjects with Gilbert's Syndrome who must have serum bilirubin < 3.0 x ULN)
13. Subject has aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) ≤ 2.5 times the ULN (OR, AST and ALT ≤ 5 times the ULN in the presence of known liver metastases)
14. Subject has alkaline phosphatase ≤ 2.5 times the ULN (OR ≤ 5 times the ULN in the presence of known liver or bone metastases)
15. Subject has normal coagulation parameters (prothrombin time [PT] and/or international normalized ratio [INR], and partial thromboplastin time [PTT] within normal limits [<1.2 x ULN])
16. Subject has potassium concentration within normal range, or correctable with supplements.
17. Oxygen saturation by pulse oximetry ≥ 92% at rest.
18. For women of childbearing potential: Negative serum pregnancy test during screening and negative serum or urine pregnancy test at start of study therapy (Cycle1 Day 1).

    Reproductive
19. For female subjects of childbearing potential, willingness to abstain from heterosexual intercourse or use a protocol-recommended method of contraception from the screening visit throughout the study treatment period and for 30 days following the last dose of study drug.
20. Female subjects of non-childbearing potential defined as having amenorrhea for at least 24 consecutive months, a documented hysterectomy, or a documented bilateral oophorectomy)
21. For fertile male subjects having intercourse with females of childbearing potential, willingness to abstain from heterosexual intercourse or use a protocol-recommended method of contraception from the start of study therapy throughout the study treatment period and for 30 days following the last dose of study drug and to refrain from sperm donation from the start of study treatment throughout the study treatment period and for 30 days following the last dose of study drug.

    Ethical
22. In the judgment of the investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the subject's cancer.
23. Before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

Disease Related

1. Subject has primary brain tumors or clinical evidence of active brain metastasis
2. Subject has undergone major surgery within 4 weeks of the start of study treatment. Laparoscopy and central venous catheter placement are not considered major surgery

   Medications
3. Subject has a history of systemic corticosteroid use within 7 days before Day 1 of Cycle 1

   General
4. Subject has an active infection requiring parenteral or oral antibiotics within 2 weeks before planned start of study therapy
5. Subject has uncontrolled diabetes as assessed by the investigator
6. Subject has a second malignancy other than curatively resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or other cancers treated with curative intent and no known active disease within 3 years before planned start of study therapy
7. Subject has an active infection of hepatitis B, hepatitis C or human immunodeficiency virus
8. Female subjects who are pregnant, planning a pregnancy or breast feeding during the study
9. Subject has a high cardiovascular risk, including, but not limited to, subjects with congestive heart failure (New York Heart Association [NYHA] Class III or IV), cardiac arrhythmia, unstable angina, coronary stenting or acute coronary syndromes within 6 months before planned start of study therapy or r myocardial infarction within one year before planned start of study therapy
10. Criterion removed
11. Subject has a history of prior allogeneic bone marrow progenitor cell or solid organ transplantation.
12. Subject has known acute or chronic pancreatitis.
13. Subject has persistent diarrhea, malabsorption, or known sub-acute bowel obstruction ≥ NCI CTCAE Grade 2, despite medical management.
14. Subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery and bariatric surgery)
15. All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before the start of study therapy (with the exception of alopecia [Grade 1 or 2 permitted], or neurotoxicity [Grade 1 or 2 permitted], or anemia [Grade 2 permitted])
16. Subject has any other medical, psychiatric, or social condition, which in the opinion of the investigator, would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results
17. Subject has a history of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies. Any lung disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
18. Subject is currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug.
19. Subject has a history of hypersensitivity to RX-3117, gemcitabine, azacytidine cytosine arabinoside, paclitaxel, nab-paclitaxel, or their excipients.
20. Subject is unwilling or unable to comply with study requirements or planned unavailability for follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ely Benaim, MD, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - Rexahn Site, Tucson, Arizona
  - Rexahn Site, Weeki Wachee, Florida
  - Rexahn Site, Joliet, Illinois
  - Rexahn Site, Skokie, Illinois
  - Rexahn Site, Lexington, Kentucky
  - Rexahn Site, Boston, Massachusetts
  - Rexahn Site, New York, New York
  - Rexahn Site, Spartanburg, South Carolina
  - Rexahn Site, Spokane, Washington
  - Rexahn Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1: The arm was designed as a dose de-escalation. De-escalation was not required during Phase 1, therefore, the starting dose 700mg RX-3117 + 125 mg/m^2 Abraxane was the only dose tested.
Groups:
- RX-3117 + Abraxane Phase 1: RX-3117: oral, 700/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once per week for 3 weeks. 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
- RX-3117 + Abraxane Phase 2: RX-3117: oral, 700 mg/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once per week for 3 weeks. 1 washout week/ cycle. (MTD)
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
Period: Overall Study
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Started | 8 | 38
Completed Cycle 1 | 6 | 31
Completed | 1 | 4
Not Completed | 7 | 34

BASELINE CHARACTERISTICS:
Groups:
- RX-3117 + Abraxane Phase 1; RX-3117 + Abraxane Phase 2: RX-3117: oral, 700 mg/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once per week for 3 weeks. 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
- Total: Total of all reporting groups
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2 | Total
Number analyzed (Participants) | 8 | 38 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (70.5) | 66.3 (66) | 66.3 (67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 19 | 24
  Male | 3 | 19 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 7 | 32 | 39
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 8 | 34 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 38 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 (Phase 1 and 2)
Description: Number of participants who experienced a treatment-related adverse event
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- RX-3117 + Abraxane Phase 1; RX-3117 + Abraxane Phase 2: RX-3117: oral, 700 mg/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once a week for 3 weeks (Days 1, 8, and 15). 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 38
Participants | 8 | 38

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Phase 1 and 2)
Description: Participants with adverse events coded using the MedDRA Dictionary (Version 20.0) to Investigations. Due to the underlying disease, not all abnormal labs are reported.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 38
Participants | 4 | 18

3. Primary Outcome: Number of Participants With Vital Sign Abnormalities (Phase 1 and 2)
Description: Number of participants with clinically significant vital sign abnormalities (Phase 1 and 2) including heart rate, respiration rate, and blood pressure
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 38
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities (Phase 1 and 2)
Description: Number of participants with clinically significant ECG abnormalities (Phase 1 and 2)
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 38
Participants | 0 | 0

5. Primary Outcome: Number of Dose-limiting Toxicities (DLTs) (Phase 1)
Time Frame: 4 weeks
Population: Phase 1 participants receiving at least 10 doses in Cycle 1 and eligible for DLT evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- RX-3117 + Abraxane: RX-3117: oral, 700 mg/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once a week for 3 weeks (Days 1, 8, and 15). 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
Arm/Group | RX-3117 + Abraxane
Number analyzed (Participants) | 6
Participants | 0

6. Primary Outcome: Number of Participants With Progression Free Survival (PFS) and/or Objective Clinical Response (Phase 2)
Description: Participants must have progression Free Survival (PFS) > 4 months or objective clinical response (complete or partial response).
Time Frame: 9 months
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 33
Participants | 17

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of RX-3117 (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Day 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Population: Pharmacokinetic sampling only performed in Phase 1 and Stage 1 of Phase 2. Twelve patients were dosed as a part of Stage 1.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
ng*hr/mL | 10500 (6490) | 8780 (4460)

8. Secondary Outcome: Time to Maximum Observed Concentration [Tmax] of RX-3117 (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Days 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
hr | 2.3 (0.89) | 4.51 (6.18)

9. Secondary Outcome: Maximum Observed Concentration [Cmax] of RX-3117 (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Days 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
ng/mL | 1120 (516) | 947 (422)

10. Secondary Outcome: Overall Response Rate [ORR] (Phase 1 and Phase 2)
Description: Overall Response Rate will be based on the RECIST v1.1 and is defined as the percentage of subjects meeting criteria of Complete Response (CR) or Partial Response (PR). CR or PR must be confirmed at least 4 weeks after the date of the original CR or PR.
Time Frame: Every 8 weeks until progression or discontinuation, whichever came first, assessed up to 32 weeks
Population: The overall number of participants analyzed is based on the modified intent-to-treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 33
Participants | 2 | 7

11. Secondary Outcome: Time to Response [TTR] (Phase 1)
Time Frame: Up to 32 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RX-3117 + Abraxane Phase 1
Number analyzed (Participants) | 6
weeks | 23.6 [7.4 to 23.6]

12. Secondary Outcome: Duration of Response [DOR] (Phase 1 and Phase 2)
Description: Duration of response is defined as the time from documentation of response to disease progression.
Time Frame: Up to 32 weeks
Population: Duration of Response was not evaluable
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- RX-3117 + Abraxane Phase 2: RX-3117: oral, 700/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once a week for 3 weeks (Days 1, 8, and 15). 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 33
weeks | NA [19.1 to NA] — The small number of patients is insufficient to calculate the median duration of response | NA [16.1 to NA] — The small number of patients is insufficient to calculate the median duration of response

13. Secondary Outcome: Progression-free Survival [PFS] (Phase 1)
Description: Progression Free Survival defined as the percentage of subjects who are alive in the study and not in progression.
Time Frame: Every 8 weeks until progression or discontinuation, whichever came first, assessed up to 32 weeks
Population: The overall number of participants analyzed is based on the modified intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- RX-3117 + Abraxane Phase 2: RX-3117: oral, 500/ day for 5 days on/ 2 days off for 3 weeks. 1 washout week/ cycle.
  Abraxane: 125 mg/m^2, infused once per week for 3 weeks. 1 washout week/ cycle.
  RX-3117: RX-3117 will be administered orally in combination with Abraxane.
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 33
weeks | 13.8 [7.0 to NA] — The value is not available because the data set is small and the upper limit of the confidence interval is non-evaluable. | 23.3 [15.1 to 31.1]

14. Secondary Outcome: Time to Progression (Phase 2)
Description: Time to Progression defined as the time from first treatment administration to first documentation of RECIST-defined objective tumor progression.
Time Frame: Every 8 weeks until progression or discontinuation, whichever came first, assessed up to 32 weeks
Population: The overall number of participants analyzed is based on the modified intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 33
weeks | 13.8 [7.0 to NA] — The value is not available because the data set is small and the upper limit of the confidence interval is non-evaluable. | 23.4 [15.1 to 32.6]

15. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of RX-3117 and Abraxane® (Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 9
ng*hr/mL | 1820 (510) | 3160 (1490)

16. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Abraxane® (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Day 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
ng*hr/mL | 5560 (2410) | 5290 (2120)

17. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Abraxane®(Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 5 | 8
ng*hr/mL | 4020 (1710) | 3670 (2080)

18. Secondary Outcome: Time to Maximum Observed Concentration [Tmax] of RX-3117 (Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 9
hr | 1.84 (0.41) | 3.75 (1.35)

19. Secondary Outcome: Time to Maximum Observed Concentration [Tmax] of Abraxane® (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Days 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
hr | 0.71 (0.17) | 0.62 (0.10)

20. Secondary Outcome: Time to Maximum Observed Concentration [Tmax] of Abraxane® (Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 5 | 8
hr | 0.55 (0.06) | 0.69 (0.18)

21. Other Pre Specified Outcome: Exploratory Measurement of Protein Biomarkers Related to RX-3117 or Pancreatic Cancer (Phase 1 and 2)
Time Frame: Baseline, and at 8, 6, 24, and 32 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Tumor Burden Response (Phase 2)
Description: Changes in tumor burden response via tumor marker measurement
Time Frame: Baseline, and at 8, 6, 24, and 32 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Quality of Life (QOL) (Phase 1 and 2)
Description: Weekly patient reported quality of life measures using validated QOL questionnaires
Time Frame: 9 months
Reporting Status: Not Posted

24. Secondary Outcome: Maximum Observed Concentration [Cmax] of RX-3117 (Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 6 | 9
ng/mL | 528 (166) | 838 (329)

25. Secondary Outcome: Maximum Observed Concentration [Cmax] of Abraxane (Phase 1 and Phase 2) - Day 1
Time Frame: Cycle 1 Days 1 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, 6, and 24 hours after administration)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 8 | 12
ng/mL | 4160 (2770) | 3940 (2320)

26. Secondary Outcome: Maximum Observed Concentration [Cmax] of Abraxane (Phase 1 and Phase 2) - Day 15
Time Frame: Day 15 (pre-infusion, post-infusion, pre-dose RX-3117, and 0.5, 1, 2, 4, and 6 hours after administration)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
Number analyzed (Participants) | 5 | 8
ng/mL | 4780 (2380) | 3320 (2330)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Cycle 1 Day until Safety Follow Up (30 days after last dose). an average of 9 months.
Arm/Group | RX-3117 + Abraxane Phase 1 | RX-3117 + Abraxane Phase 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 2/38
Serious Adverse Events (participants affected / at risk) | 3/8 | 18/38
Other Adverse Events (participants affected / at risk) | 8/8 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RX-3117 + Abraxane Phase 1 (N=8) | RX-3117 + Abraxane Phase 2 (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Emphysematous choleccystitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Penumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musucular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RX-3117 + Abraxane Phase 1 (N=8) | RX-3117 + Abraxane Phase 2 (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 | 19
Neutropenia (Blood and lymphatic system disorders) | 1 | 9
Palpitations (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 25
Nausea (Gastrointestinal disorders) | 6 | 23
Abdominal pain (Gastrointestinal disorders) | 1 | 20
Vomiting (Gastrointestinal disorders) | 4 | 11
Constipation (Gastrointestinal disorders) | 2 | 12
Abdominal distension (Gastrointestinal disorders) | 0 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Flatulence (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Fatigue (Gastrointestinal disorders) | 6 | 23
Pyrexia (Gastrointestinal disorders) | 2 | 13
Oedema peripheral (Gastrointestinal disorders) | 1 | 13
Chills (Gastrointestinal disorders) | 1 | 7
Asthenia (Gastrointestinal disorders) | 2 | 5
Non-cardiac chest pain (Gastrointestinal disorders) | 0 | 5
Influenza like illness (Gastrointestinal disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 5
Oral candidiasis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 3
Weight decreased (Investigations) | 0 | 7
Blood bilirubin increased (Investigations) | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Neutrophil count decreased (Investigations) | 1 | 4
White blood cell count decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 15
Dehydration (Metabolism and nutrition disorders) | 2 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 2 | 17
Neuropathy peripheral (Nervous system disorders) | 1 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 8
Dysgeusia (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 2 | 5
Depression (Psychiatric disorders) | 0 | 7
Insomnia (Psychiatric disorders) | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9
Rash (Skin and subcutaneous tissue disorders) | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03189914/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03189914/SAP_001.pdf